CLINICAL TRIAL: NCT01106651
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Multicenter Study to Evaluate the Efficacy, Safety, and Tolerability of Canagliflozin Compared With Placebo in the Treatment of Older Subjects With Type 2 Diabetes Mellitus Inadequately Controlled on Glucose Lowering Therapy
Brief Title: A Safety and Efficacy Study of Canagliflozin in Older Patients (55 to 80 Years of Age) With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CR017014; 28431754DIA3010 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2010-04-01; First posted 2010-04-20 (Estimated); Results first posted 2013-05-29 (Estimated); Last update posted 2014-11-04 (Estimated); Status verified 2014-10

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Canagliflozin; Placebo; Hemoglobin A1c; Bone; Type 2 diabetes mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Canagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Canagliflozin 100 mg (Experimental): Each patient will receive 100 mg of canagliflozin once daily for 104 weeks with/without stable doses of antihyperglycemic agent(s) taken at the time of study entry.
  Interventions: Drug: Canagliflozin 100 mg; Drug: Antihyperglycemic agent(s)
- Canagliflozin 300 mg (Experimental): Each patient will receive 300 mg of canagliflozin once daily for 104 weeks with/without stable doses of antihyperglycemic agent(s) taken at the time of study entry.
  Interventions: Drug: Canagliflozin 300 mg; Drug: Antihyperglycemic agent(s)
- Placebo (Placebo Comparator): Each patient will receive matching placebo once daily for 104 weeks with/without stable doses of antihyperglycemic agent(s) taken at the time of study entry.
  Interventions: Drug: Antihyperglycemic agent(s); Drug: Placebo

INTERVENTIONS:
Drug: Canagliflozin 100 mg — One 100 mg over-encapsulated tablet orally (by mouth) once daily for 104 weeks with/without stable doses of antihyperglycemic agent(s) taken at the time of study entry.
  Arms: Canagliflozin 100 mg
Drug: Canagliflozin 300 mg — One 300 mg over-encapsulated tablet orally (by mouth) once daily for 104 weeks with/without stable doses of antihyperglycemic agent(s) taken at the time of study entry.
  Arms: Canagliflozin 300 mg
Drug: Antihyperglycemic agent(s) — Stable doses of antihyperglycemic agents (sulfonylurea agent, thiazolidinediones, dipeptidyl peptidase 4 [DPP-4] inhibitors, metformin, insulin [all types]) and their combinations (sulfonylurea agent and insulin [all types], metformin and insulin [all types], metformin and sulfonylurea, alpha glucosidase inhibitors, thiazolidinediones, dipeptidyl peptidase 4 [DPP-4]) are used as per protocol specifications.
Drug: Placebo — One matching placebo capsule orally once daily for 104 weeks with/without stable doses of antihyperglycemic agent(s) taken at the time of study entry.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of 2 different doses of canagliflozin compared with placebo in older patients (55 to 80 years of age) with type 2 diabetes mellitus (T2DM) with inadequate control on their current diabetes treatment regimen.

DETAILED DESCRIPTION:
Canagliflozin is a drug that is being tested to see if it may be useful in treating patients diagnosed with type 2 diabetes mellitus (T2DM). This is a randomized (study drug assigned by chance), double-blind (neither the patient or the study doctor will know the name of the assigned treatment), placebo-controlled, parallel-group, 3-arm (3 treatment groups) multicenter study to determine the efficacy, safety, and tolerability of canagliflozin (100 mg and 300 mg) compared to placebo (a capsule that looks like all the other treatments but has no real medicine) in patients with T2DM who are not achieving an adequate response from current antihyperglycemic therapy to control their diabetes. Approximately 720 older (55 to 80 years of age) patients with T2DM who are either not on an antihyperglycemic agent or who are receiving treatment with a stable regimen of antihyperglycemic agent(s) and have inadequate glycemic (blood sugar) control will receive once daily treatment with canagliflozin (100 mg or 300 mg) or placebo capsules for 104 weeks (includes 26 weeks of double-blind treatment followed by a 78-week extension period). In addition, all patients will take stable doses of the antihyperglycemic agent(s) that they were taking before entry in the study for the duration of the study. Patients will participate in the study for approximately 108 weeks. During the study, if a patient's fasting blood sugar remains high despite treatment with study drug, the patient will receive treatment with an antihyperglycemic agent (rescue therapy) that is considered clinically appropriate and consistent with local prescribing information. During treatment, patients will be monitored for safety by review of adverse events, results from laboratory tests, measures of bone health, 12-lead electrocardiograms (ECGs), vital signs measurements, body weight, physical examinations, and self-monitored blood glucose (SMGB) measurements. The primary outcome measure in the study is the effect of canagliflozin relative to placebo on hemoglobin A1c (HbA1c) after 26 weeks of treatment. Study drug will be taken orally (by mouth) once daily before the first meal each day unless otherwise specified. All patients will take single-blind placebo capsules for 2 weeks before randomization. After randomization, patients will take double blind canagliflozin (100 mg or 300 mg) or matching placebo for 104 weeks.

ELIGIBILITY:
Inclusion Criteria:

* All patients must have a diagnosis of T2DM and may be currently treated with a stable regimen of antihyperglycemic agent(s)
* Patients in the study must have a HbA1c between >=7 and <=10.0%
* Patients must have a fasting plasma glucose (FPG) <270 mg/dL (15 mmol/L)

Exclusion Criteria:

* History of diabetic ketoacidosis, type 1 diabetes mellitus (T1DM), pancreas or beta cell transplantation, or diabetes secondary to pancreatitis or pancreatectomy, or a severe hypoglycemic episode within 6 months before screening

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 716 (Actual)
Dates: Start 2010-06; Primary Completion 2011-11 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (86):
- United States (34):
  - Glendale, Arizona
  - Phoenix, Arizona
  - Little Rock, Arkansas
  - Carmichael, California
  - Citrus Heights, California
  - Fair Oaks, California
  - Roseville, California
  - Sacramento, California
  - San Diego, California
  - Walnut Creek, California
  - Daytona Beach, Florida
  - Fleming Island, Florida
  - Jacksonville, Florida
  - Miami, Florida
  - Atlanta, Georgia
  - Wichita, Kansas
  - Waltham, Massachusetts
  - Pahrump, Nevada
  - Albuquerque, New Mexico
  - Cary, North Carolina
  - Charlotte, North Carolina
  - Wilmington, North Carolina
  - Bismarck, North Dakota
  - Franklin, Ohio
  - Mt. Pleasant, South Carolina
  - Bristol, Tennessee
  - Carrollton, Texas
  - Dallas, Texas
  - Irving, Texas
  - Plano, Texas
  - Richardson, Texas
  - Renton, Washington
  - Tacoma, Washington
  - Wenatchee, Washington
- Australia (4):
  - Fremantle
  - Heidelberg Heights
  - Meadowbrook
  - Richmond
- Canada (8):
  - Vancouver, British Columbia
  - St. John's, Newfoundland and Labrador
  - Barrie, Ontario
  - London, Ontario
  - Markham, Ontario
  - Oakville, Ontario
  - Toronto, Ontario
  - Montreal, Quebec
- Colombia (2):
  - Barranquilla
  - Bogotá
- France (3):
  - Corbeil-Essonnes
  - Paris
  - Vénissieux
- Greece (2):
  - Thessaloniki
  - Thessalonikis
- Shatin, Hong Kong
- India (3):
  - Bangalore
  - Nagpur
  - Pune
- New Zealand (4):
  - Auckland
  - Christchurch
  - Tauranga
  - Wellington
- Poland (5):
  - Katowice
  - Krakow
  - Torun
  - Warsaw
  - Wroclaw
- Romania (2):
  - Bucharest
  - Sibiu
- Pretoria, South Africa
- Spain (4):
  - Granada
  - Madrid
  - Pozuelo de Alarcón
  - Seville
- Sweden (2):
  - Gothenburg
  - Uppsala
- Switzerland (2):
  - Bruderholz
  - Sankt Gallen
- Ukraine (2):
  - Kharkiv
  - Kiev
- United Kingdom (7):
  - Birmingham
  - Cardiff
  - Glasgow
  - Liverpool
  - Manchester
  - Reading
  - Salford

REFERENCES:
- [Derived] Januzzi JL Jr, Butler J, Jarolim P, Sattar N, Vijapurkar U, Desai M, Davies MJ. Effects of Canagliflozin on Cardiovascular Biomarkers in Older Adults With Type 2 Diabetes. J Am Coll Cardiol. 2017 Aug 8;70(6):704-712. doi: 10.1016/j.jacc.2017.06.016. Epub 2017 Jun 12. PMID 28619659
- [Derived] Qiu R, Balis D, Xie J, Davies MJ, Desai M, Meininger G. Longer-term safety and tolerability of canagliflozin in patients with type 2 diabetes: a pooled analysis. Curr Med Res Opin. 2017 Mar;33(3):553-562. doi: 10.1080/03007995.2016.1271780. Epub 2017 Jan 4. PMID 27977934
- [Derived] Blonde L, Stenlof K, Fung A, Xie J, Canovatchel W, Meininger G. Effects of canagliflozin on body weight and body composition in patients with type 2 diabetes over 104 weeks. Postgrad Med. 2016 May;128(4):371-80. doi: 10.1080/00325481.2016.1169894. Epub 2016 Apr 7. PMID 27002421
- [Derived] Watts NB, Bilezikian JP, Usiskin K, Edwards R, Desai M, Law G, Meininger G. Effects of Canagliflozin on Fracture Risk in Patients With Type 2 Diabetes Mellitus. J Clin Endocrinol Metab. 2016 Jan;101(1):157-66. doi: 10.1210/jc.2015-3167. Epub 2015 Nov 18. PMID 26580237
- [Derived] Bilezikian JP, Watts NB, Usiskin K, Polidori D, Fung A, Sullivan D, Rosenthal N. Evaluation of Bone Mineral Density and Bone Biomarkers in Patients With Type 2 Diabetes Treated With Canagliflozin. J Clin Endocrinol Metab. 2016 Jan;101(1):44-51. doi: 10.1210/jc.2015-1860. Epub 2015 Nov 18. PMID 26580234
- [Derived] Weir MR, Kline I, Xie J, Edwards R, Usiskin K. Effect of canagliflozin on serum electrolytes in patients with type 2 diabetes in relation to estimated glomerular filtration rate (eGFR). Curr Med Res Opin. 2014 Sep;30(9):1759-68. doi: 10.1185/03007995.2014.919907. Epub 2014 May 22. PMID 24786834
- [Derived] Nyirjesy P, Sobel JD, Fung A, Mayer C, Capuano G, Ways K, Usiskin K. Genital mycotic infections with canagliflozin, a sodium glucose co-transporter 2 inhibitor, in patients with type 2 diabetes mellitus: a pooled analysis of clinical studies. Curr Med Res Opin. 2014 Jun;30(6):1109-19. doi: 10.1185/03007995.2014.890925. Epub 2014 Feb 21. PMID 24517339
- [Derived] Bode B, Stenlof K, Sullivan D, Fung A, Usiskin K. Efficacy and safety of canagliflozin treatment in older subjects with type 2 diabetes mellitus: a randomized trial. Hosp Pract (1995). 2013 Apr;41(2):72-84. doi: 10.3810/hp.2013.04.1020. PMID 23680739

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study evaluated the efficacy and safety of canagliflozin in older patients with type 2 diabetes mellitus with inadequate control on their current diabetes treatment regimen. The study began on 07 June 2010 and ended on 23 May 2013. Patients were recruited from 90 study centers located in 17 countries worldwide.
Pre-assignment Details: 716 patients were randomly allocated to the 3 treatment arms. 714 patients received at least 1 dose of study drug and were included in the modified intent-to-treat (mITT) analysis set and safety analysis set. Participant flow is presented for Baseline to Week 104 (Overall Study).
Groups:
- Placebo: Each patient received matching placebo once daily for 104 weeks in addition to being on a stable antihyperglycemic (AHA) regimen at the time of study entry.
- Canagliflozin 100 mg: Each patient received 100 mg of canagliflozin once daily for 104 weeks in addition to being on a stable antihyperglycemic (AHA) regimen at the time of study entry.
- Canagliflozin 300 mg: Each patient received 300 mg of canagliflozin once daily for 104 weeks in addition to being on a stable antihyperglycemic (AHA) regimen at the time of study entry.
Period: Overall Study
Arm/Group | Placebo | Canagliflozin 100 mg | Canagliflozin 300 mg
Started | 237 | 241 | 236
Completed | 158 | 184 | 178
Not Completed | 79 | 57 | 58
Not completed — Adverse Event | 17 | 9 | 23
Not completed — Lost to Follow-up | 8 | 2 | 6
Not completed — Physician Decision | 4 | 3 | 1
Not completed — Protocol Violation | 1 | 2 | 1
Not completed — Withdrawal by Subject | 14 | 7 | 4
Not completed — Noncompliance with study drug | 1 | 0 | 2
Not completed — Other | 34 | 31 | 21
Not completed — Death | 0 | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Canagliflozin 100 mg | Canagliflozin 300 mg | Total
Number analyzed (Participants) | 237 | 241 | 236 | 714
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 151 | 141 | 149 | 441
  >=65 years | 86 | 100 | 87 | 273
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.2 (6.21) | 64.3 (6.46) | 63.4 (5.99) | 63.6 (6.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 94 | 117 | 107 | 318
  Male | 143 | 124 | 129 | 396
Region of Enrollment [Number; unit: participants]
  AUSTRALIA | 6 | 6 | 11 | 23
  CANADA | 24 | 32 | 28 | 84
  COLOMBIA | 18 | 15 | 20 | 53
  FRANCE | 2 | 2 | 3 | 7
  GREECE | 1 | 1 | 1 | 3
  HONG KONG | 1 | 1 | 2 | 4
  INDIA | 8 | 3 | 11 | 22
  NEW ZEALAND | 16 | 10 | 11 | 37
  POLAND | 11 | 12 | 14 | 37
  ROMANIA | 8 | 10 | 7 | 25
  SOUTH AFRICA | 9 | 12 | 10 | 31
  SPAIN | 2 | 3 | 8 | 13
  SWEDEN | 4 | 4 | 2 | 10
  SWITZERLAND | 2 | 2 | 0 | 4
  UKRAINE | 3 | 8 | 3 | 14
  UNITED KINGDOM | 19 | 22 | 8 | 49
  UNITED STATES | 103 | 98 | 97 | 298

OUTCOME MEASURES:

1. Primary Outcome: Change in HbA1c From Baseline to Week 26
Description: The table below shows the least-squares (LS) mean change in HbA1c from Baseline to Week 26 for each treatment group. The statistical analyses show the treatment differences (ie, each canagliflozin group minus placebo) in the LS mean change.
Time Frame: Day 1 (Baseline) and Week 26
Population: Analysis used mITT analysis set (all randomized patients who received at least 1 dose of study drug). Last-observation-carried-forward method used for missing Week 26 values. Measurements taken pre-rescue used as last observation in patients receiving glycemic rescue therapy. Table includes only patients with both baseline and post baseline values.
Measure: Least Squares Mean (Standard Error); unit: Percent
Arm/Group | Placebo | Canagliflozin 100 mg | Canagliflozin 300 mg
Number analyzed (Participants) | 232 | 239 | 229
Percent | -0.03 (0.063) | -0.60 (0.063) | -0.73 (0.064)
Statistical Analysis 1: Comparison: Placebo vs Canagliflozin 100 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; Least-Squares Mean Difference = -0.57, 95% CI 2-sided [-0.708 to -0.436], Standard Error of Mean 0.069
Statistical Analysis 2: Comparison: Placebo vs Canagliflozin 300 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; Least-Squares Mean Difference = -0.70, 95% CI 2-sided [-0.841 to -0.566], Standard Error of Mean 0.070

2. Secondary Outcome: Percentage of Patients With HbA1c <7% at Week 26
Description: The table below shows the percentage of patients with HbA1c <7% at Week 26 in each treatment group. The statistical analyses show the treatment differences (ie, each canagliflozin group minus placebo) in the percentage.
Time Frame: Week 26
Population: as for outcome 1
Measure: Number; unit: Percentage of patients
Arm/Group | Placebo | Canagliflozin 100 mg | Canagliflozin 300 mg
Number analyzed (Participants) | 232 | 239 | 229
Percentage of patients | 28.0 | 47.7 | 58.5
Statistical Analysis 1: Comparison: Placebo vs Canagliflozin 100 mg; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 2.96, 95% CI [1.93 to 4.56]
Statistical Analysis 2: Comparison: Placebo vs Canagliflozin 300 mg; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 4.48, 95% CI [2.89 to 6.95]

3. Secondary Outcome: Change in Fasting Plasma Glucose (FPG) From Baseline to Week 26
Description: The table below shows the least-squares (LS) mean change in FPG from Baseline to Week 26 for each treatment group. The statistical analyses show the treatment differences (ie, each canagliflozin group minus placebo) in the LS mean change.
Time Frame: Day 1 (Baseline) and Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Canagliflozin 100 mg | Canagliflozin 300 mg
Number analyzed (Participants) | 231 | 239 | 229
mg/dL | 7.39 (2.875) | -18.1 (2.860) | -20.3 (2.920)
Statistical Analysis 1: Comparison: Placebo vs Canagliflozin 100 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; Least-Squares Mean Difference = -25.5, 95% CI 2-sided [-31.68 to -19.32], Standard Error of Mean 3.147
Statistical Analysis 2: Comparison: Placebo vs Canagliflozin 300 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; Least-Squares Mean Difference = -27.7, 95% CI 2-sided [-33.97 to -21.49], Standard Error of Mean 3.179

4. Secondary Outcome: Percent Change in Body Weight From Baseline to Week 26
Description: The table below shows the least-squares (LS) mean percent change in body weight from Baseline to Week 26 for each treatment group. The statistical analyses show the treatment differences (ie, each canagliflozin group minus placebo) in the LS mean change.
Time Frame: Day 1 (Baseline) and Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Placebo | Canagliflozin 100 mg | Canagliflozin 300 mg
Number analyzed (Participants) | 234 | 240 | 229
Percent change | -0.1 (0.3) | -2.4 (0.3) | -3.1 (0.3)
Statistical Analysis 1: Comparison: Placebo vs Canagliflozin 100 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; Least-Squares Mean Difference = -2.3, 95% CI 2-sided [-2.8 to -1.7], Standard Error of Mean 0.3
Statistical Analysis 2: Comparison: Placebo vs Canagliflozin 300 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; Least-Squares Mean Difference = -3.0, 95% CI 2-sided [-3.5 to -2.4], Standard Error of Mean 0.3

5. Secondary Outcome: Change in Total Fat From Baseline to Week 26 in a Subset of Patients Undergoing Specific Dual-energy X-ray Absorptiometry (DXA) Analysis for Body Composition
Description: The table below shows the least-squares (LS) mean change in total fat from Baseline to Week 26 for each treatment group in patients randomized to the subset of patients undergoing specific DXA analysis for body composition. The statistical analyses show the treatment differences (ie, each canagliflozin group minus placebo) in the LS mean change.
Time Frame: Day 1 (Baseline) and Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | Placebo | Canagliflozin 100 mg | Canagliflozin 300 mg
Number analyzed (Participants) | 50 | 56 | 60
kg | -0.28 (0.336) | -1.87 (0.332) | -2.38 (0.323)
Statistical Analysis 1: Comparison: Placebo vs Canagliflozin 100 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; Least-Squares Mean Difference = -1.59, 95% CI 2-sided [-2.339 to -0.842], Standard Error of Mean 0.379
Statistical Analysis 2: Comparison: Placebo vs Canagliflozin 300 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; Least-Squares Mean Difference = -2.10, 95% CI 2-sided [-2.833 to -1.368], Standard Error of Mean 0.371

6. Secondary Outcome: Change in Region Percent Total Fat From Baseline to Week 26 in a Subset of Patients Undergoing Specific Dual-energy X-ray Absorptiometry (DXA) Analysis for Body Composition
Description: Region percent total fat = body fat as a percentage of (body fat + lean body mass + bone mass content). The table below shows the least-squares (LS) mean change in region percent total fat from Baseline to Week 26 for each treatment group in patients randomized to the subset of patients undergoing specific dual-energy X-ray absorptiometry (DXA) analysis for body composition. The statistical analyses show the treatment differences (ie, each canagliflozin group minus placebo) in the LS mean change.
Time Frame: Day 1 (Baseline) and Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Percent
Arm/Group | Placebo | Canagliflozin 100 mg | Canagliflozin 300 mg
Number analyzed (Participants) | 50 | 56 | 60
Percent | 0.00 (0.270) | -1.03 (0.268) | -1.18 (0.261)
Statistical Analysis 1: Comparison: Placebo vs Canagliflozin 100 mg; Region percent total fat; Test type: Superiority or Other; p < 0.001, ANCOVA; Least-Squares Mean Difference = -1.03, 95% CI 2-sided [-1.633 to -0.428], Standard Error of Mean 0.305
Statistical Analysis 2: Comparison: Placebo vs Canagliflozin 300 mg; Region percent total fat; Test type: Superiority or Other; p < 0.001, ANCOVA; Least-Squares Mean Difference = -1.18, 95% CI 2-sided [-1.772 to -0.587], Standard Error of Mean 0.300

7. Secondary Outcome: Change in Tissue Percent Total Fat From Baseline to Week 26 in a Subset of Patients Undergoing Specific Dual-energy X-ray Absorptiometry (DXA) Analysis for Body Composition
Description: Tissue percent total fat = body fat as a percentage of body fat + lean body mass. The table below shows the least-squares (LS) mean change in tissue percent total fat from Baseline to Week 26 for each treatment group in patients randomized to the subset of patients undergoing specific DXA analysis for body composition. The statistical analyses show the treatment differences (ie, each canagliflozin group minus placebo) in the LS mean change.
Time Frame: Day 1 (Baseline) and Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Percent
Arm/Group | Placebo | Canagliflozin 100 mg | Canagliflozin 300 mg
Number analyzed (Participants) | 50 | 56 | 60
Percent | 0.02 (0.280) | -1.04 (0.278) | -1.18 (0.270)
Statistical Analysis 1: Comparison: Placebo vs Canagliflozin 100 mg; Test type: Superiority or Other; p = 0.001, ANCOVA; Least-Squares Mean Difference = -1.05, 95% CI 2-sided [-1.677 to -0.430], Standard Error of Mean 0.316
Statistical Analysis 2: Comparison: Placebo vs Canagliflozin 300 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; Least-Squares Mean Difference = -1.20, 95% CI 2-sided [-1.812 to -0.584], Standard Error of Mean 0.311

8. Secondary Outcome: Change in Systolic Blood Pressure (SBP) From Baseline to Week 26
Description: The table below shows the least-squares (LS) mean change in SBP from Baseline to Week 26 for each treatment group. The statistical analyses show the treatment differences (ie, each canagliflozin group minus placebo) in the LS mean change.
Time Frame: Day 1 (Baseline) and Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Placebo | Canagliflozin 100 mg | Canagliflozin 300 mg
Number analyzed (Participants) | 234 | 240 | 229
mmHg | 1.10 (1.039) | -3.52 (1.035) | -6.79 (1.056)
Statistical Analysis 1: Comparison: Placebo vs Canagliflozin 100 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; Least-Squares Mean Difference = -4.63, 95% CI 2-sided [-6.854 to -2.401], Standard Error of Mean 1.134
Statistical Analysis 2: Comparison: Placebo vs Canagliflozin 300 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; Least-Squares Mean Difference = -7.89, 95% CI 2-sided [-10.14 to -5.641], Standard Error of Mean 1.147

9. Secondary Outcome: Percent Change in Triglycerides From Baseline to Week 26
Description: The table below shows the least-squares (LS) mean percent change in triglycerides from Baseline to Week 26 for each treatment group. The statistical analyses show the treatment differences (ie, each canagliflozin group minus placebo) in the LS mean change.
Time Frame: Day 1 (Baseline) and Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Placebo | Canagliflozin 100 mg | Canagliflozin 300 mg
Number analyzed (Participants) | 206 | 227 | 222
Percent change | 7.7 (3.4) | 2.8 (3.3) | 8.4 (3.4)
Statistical Analysis 1: Comparison: Placebo vs Canagliflozin 100 mg; Test type: Superiority or Other; p = 0.194, ANCOVA; Least-Squares Mean Difference = -4.8, 95% CI 2-sided [-12.1 to 2.5], Standard Error of Mean 3.7
Statistical Analysis 2: Comparison: Placebo vs Canagliflozin 300 mg; Test type: Superiority or Other; p = 0.846, ANCOVA; Least-Squares Mean Difference = 0.7, 95% CI 2-sided [-6.6 to 8.1], Standard Error of Mean 3.7

10. Secondary Outcome: Percent Change in High-density Lipoprotein Cholesterol (HDL-C) From Baseline to Week 26
Description: The table below shows the least-squares (LS) mean percent change in HDL-C from Baseline to Week 26 or each treatment group. The statistical analyses show the treatment differences (ie, each canagliflozin group minus placebo) in the LS mean change.
Time Frame: Day 1 (Baseline) and Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Placebo | Canagliflozin 100 mg | Canagliflozin 300 mg
Number analyzed (Participants) | 206 | 225 | 222
Percent change | 1.5 (1.2) | 6.8 (1.2) | 6.2 (1.2)
Statistical Analysis 1: Comparison: Placebo vs Canagliflozin 100 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; Least-Squares Mean Difference = 5.3, 95% CI 2-sided [2.6 to 7.9], Standard Error of Mean 1.4
Statistical Analysis 2: Comparison: Placebo vs Canagliflozin 300 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; Least-Squares Mean Difference = 4.7, 95% CI 2-sided [2.0 to 7.4], Standard Error of Mean 1.4

11. Secondary Outcome: Percent Change in Lumbar Spine Bone Mineral Density (BMD) From Baseline to Week 26
Description: The table below shows the least-squares (LS) mean percent change from Baseline to Week 26 in lumbar spine BMD for each treatment group as assessed by dual-energy X-ray absorptiometry (DXA). The statistical analyses show the treatment differences (ie, each canagliflozin group minus placebo) in LS mean percent change.
Time Frame: Day 1 (Baseline) and Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Placebo | Canagliflozin 100 mg | Canagliflozin 300 mg
Number analyzed (Participants) | 185 | 206 | 192
Percent change | 0.5 (0.3) | 0.7 (0.3) | 0.2 (0.3)
Statistical Analysis 1: Comparison: Placebo vs Canagliflozin 100 mg; Test type: Superiority or Other; ANCOVA; Least-Squares Mean Difference = 0.2, 95% CI 2-sided [-0.4 to 0.8], Standard Error of Mean 0.3
Statistical Analysis 2: Comparison: Placebo vs Canagliflozin 300 mg; Test type: Superiority or Other; ANCOVA; Least-Squares Mean Difference = -0.3, 95% CI 2-sided [-0.9 to 0.3], Standard Error of Mean 0.3

12. Secondary Outcome: Percent Change in Distal Forearm Bone Mineral Density (BMD) From Baseline to Week 26
Description: The table below shows the least-squares (LS) mean percent change from Baseline to Week 26 in distal forearm BMD for each treatment group as assessed by dual-energy X-ray absorptiometry (DXA). The statistical analyses show the treatment differences (ie, each canagliflozin group minus placebo) in LS mean percent change.
Time Frame: Day 1 (Baseline) and Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Placebo | Canagliflozin 100 mg | Canagliflozin 300 mg
Number analyzed (Participants) | 187 | 208 | 187
Percent change | -0.5 (0.3) | -0.7 (0.3) | -0.8 (0.3)
Statistical Analysis 1: Comparison: Placebo vs Canagliflozin 100 mg; Test type: Superiority or Other; ANCOVA; Least-Squares Mean Difference = -0.3, 95% CI 2-sided [-0.9 to 0.4], Standard Error of Mean 0.3
Statistical Analysis 2: Comparison: Placebo vs Canagliflozin 300 mg; Test type: Superiority or Other; ANCOVA; Least-Squares Mean Difference = -0.4, 95% CI 2-sided [-1.0 to 0.3], Standard Error of Mean 0.3

13. Secondary Outcome: Percent Change in Femoral Neck Bone Mineral Density (BMD) From Baseline to Week 26
Description: The table below shows the least-squares (LS) mean percent change from Baseline to Week 26 in femoral neck BMD for each treatment group as assessed by dual-energy X-ray absorptiometry (DXA). The statistical analyses show the treatment differences (ie, each canagliflozin group minus placebo) in LS mean percent change.
Time Frame: Day 1 (Baseline) and Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Placebo | Canagliflozin 100 mg | Canagliflozin 300 mg
Number analyzed (Participants) | 183 | 209 | 190
Percent change | -1.0 (0.3) | -0.7 (0.3) | -0.6 (0.3)
Statistical Analysis 1: Comparison: Placebo vs Canagliflozin 100 mg; Test type: Superiority or Other; ANCOVA; Least-Squares Mean Difference = 0.3, 95% CI 2-sided [-0.3 to 1.0], Standard Error of Mean 0.3
Statistical Analysis 2: Comparison: Placebo vs Canagliflozin 300 mg; Test type: Superiority or Other; ANCOVA; Least-Squares Mean Difference = 0.4, 95% CI 2-sided [-0.3 to 1.1], Standard Error of Mean 0.3

14. Secondary Outcome: Percent Change in Total Hip Bone Mineral Density (BMD) From Baseline to Week 26
Description: The table below shows the least-squares (LS) mean percent change from Baseline to Week 26 in total hip BMD for each treatment group as assessed by dual-energy X-ray absorptiometry (DXA). The statistical analyses show the treatment differences (ie, each canagliflozin group minus placebo) in LS mean percent change.
Time Frame: Day 1 (Baseline) and Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Placebo | Canagliflozin 100 mg | Canagliflozin 300 mg
Number analyzed (Participants) | 183 | 209 | 190
Percent change | -0.5 (0.2) | -0.9 (0.2) | -1.0 (0.2)
Statistical Analysis 1: Comparison: Placebo vs Canagliflozin 100 mg; Test type: Superiority or Other; ANCOVA; Least-Squares Mean Difference = -0.4, 95% CI 2-sided [-0.8 to -0.0], Standard Error of Mean 0.2
Statistical Analysis 2: Comparison: Placebo vs Canagliflozin 300 mg; Test type: Superiority or Other; ANCOVA; Least-Squares Mean Difference = -0.5, 95% CI 2-sided [-0.9 to -0.1], Standard Error of Mean 0.2

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for the duration of the study (104 weeks).
Description: The total number of adverse events listed in the "Other (non-Serious) Adverse Events" table are based upon a cut-off of greater than or equal to 5 percent of patients experiencing the adverse event in any treatment arm. MEDDRA 14.0 used for Week 26 results/ MEDDRA 16.0 used for Week 104 results.
Groups:
- Placebo: Baseline to Week 26: Each patient received matching placebo once daily for 104 weeks in addition to being on a stable antihyperglycemic (AHA) regimen at the time of study entry. Data are presented for Baseline to Week 26.
- Canagliflozin 100 mg: Baseline to Week 26: Each patient received 100 mg of canagliflozin once daily for 104 weeks in addition to being on a stable antihyperglycemic (AHA) regimen at the time of study entry. Data are presented for Baseline to Week 26.
- Canagliflozin 300 mg: Baseline to Week 26: Each patient received 300 mg of canagliflozin once daily for 104 weeks in addition to being on a stable antihyperglycemic (AHA) regimen at the time of study entry. Data are presented for Baseline to Week 26.
- Placebo: Baseline to Week 104: Each patient received matching placebo once daily for 104 weeks in addition to being on a stable antihyperglycemic (AHA) regimen at the time of study entry. Data are presented for Baseline to Week 104.
- Canagliflozin 100 mg: Baseline to Week 104: Each patient received 100 mg of canagliflozin once daily for 104 weeks in addition to being on a stable antihyperglycemic (AHA) regimen at the time of study entry. Data are presented for Baseline to Week 104
- Canagliflozin 300 mg: Baseline to Week 104: Each patient received 300 mg of canagliflozin once daily for 104 weeks in addition to being on a stable antihyperglycemic (AHA) regimen at the time of study entry. Data are presented for Baseline to Week 104
Arm/Group | Placebo: Baseline to Week 26 | Canagliflozin 100 mg: Baseline to Week 26 | Canagliflozin 300 mg: Baseline to Week 26 | Placebo: Baseline to Week 104 | Canagliflozin 100 mg: Baseline to Week 104 | Canagliflozin 300 mg: Baseline to Week 104
Serious Adverse Events (participants affected / at risk) | 12/237 | 10/241 | 8/236 | 41/237 | 40/241 | 43/236
Other Adverse Events (participants affected / at risk) | 99/237 | 92/241 | 98/236 | 166/237 | 169/241 | 169/236
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo: Baseline to Week 26 (N=237) | Canagliflozin 100 mg: Baseline to Week 26 (N=241) | Canagliflozin 300 mg: Baseline to Week 26 (N=236) | Placebo: Baseline to Week 104 (N=237) | Canagliflozin 100 mg: Baseline to Week 104 (N=241) | Canagliflozin 300 mg: Baseline to Week 104 (N=236)
Angina pectoris (Cardiac disorders) | 0 | 1 | 0 | 1 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0 | 2 | 1 | 3
Bradycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 1
Coronary artery disease (Cardiac disorders) | 1 | 0 | 0 | 3 | 3 | 3
Myocardial infarction (Cardiac disorders) | 2 | 0 | 1 | 2 | 1 | 2
Myocarditis (Cardiac disorders) | 1 | 0 | 0 | 1 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1
Intestinal infarction (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0
Umbilical hernia, obstructive (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 2 | 2 | 0 | 3
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 1 | 1 | 0
Urosepsis (Infections and infestations) | 2 | 0 | 0 | 2 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 2 | 0
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 1 | 2
Bronchioloalveolar carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 2 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 1 | 0
Carotid artery stenosis (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 0 | 0 | 3 | 1
Presyncope (Nervous system disorders) | 0 | 1 | 0 | 0 | 1 | 0
Post-traumatic stress disorder (Psychiatric disorders) | 0 | 1 | 0 | 0 | 1 | 0
Renal colic (Renal and urinary disorders) | 1 | 0 | 0 | 2 | 0 | 0
Renal impairment (Renal and urinary disorders) | 1 | 0 | 1 | 1 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 2 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1 | 0
Diplopia (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 2
Angina unstable (Cardiac disorders) | 0 | 0 | 0 | 2 | 0 | 2
Intracardiac thrombus (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Sick sinus syndrome (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Abdominal hernia obstructive (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Gastrointestinal angiodysplasia haemorrhagic (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Inguinal hernia, obstructive (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pouchitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 2 | 1 | 0
Bile duct obstruction (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Appendicitis perforated (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Cholecystitis infective (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Otitis media (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1
Subcutaneous abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Hand fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Muscle rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Blood pressure increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Cartilage atrophy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Adrenal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Angiosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Benign salivary gland neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 2
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 2
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Cauda equina syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hepatic encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hypoglycaemic coma (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hypoglycaemic seizure (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Loss of consciousness (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Migraine with aura (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Calculus ureteric (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 3 | 1
Balanoposthitis (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1
Genital prolapse (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hypoventilation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Sinus polyp (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0
Embolism arterial (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1
Peripheral vascular disorder (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo: Baseline to Week 26 (N=237) | Canagliflozin 100 mg: Baseline to Week 26 (N=241) | Canagliflozin 300 mg: Baseline to Week 26 (N=236) | Placebo: Baseline to Week 104 (N=237) | Canagliflozin 100 mg: Baseline to Week 104 (N=241) | Canagliflozin 300 mg: Baseline to Week 104 (N=236)
Diarrhoea (Gastrointestinal disorders) | 14 | 10 | 11 | 24 | 14 | 24
Influenza (Infections and infestations) | 5 | 14 | 9 | 18 | 25 | 18
Nasopharyngitis (Infections and infestations) | 19 | 23 | 19 | 36 | 45 | 44
Upper respiratory tract infection (Infections and infestations) | 11 | 13 | 10 | 29 | 23 | 25
Urinary tract infection (Infections and infestations) | 9 | 14 | 17 | 21 | 32 | 35
Hypoglycaemia (Metabolism and nutrition disorders) | 34 | 25 | 23 | 47 | 37 | 36
Arthralgia (Musculoskeletal and connective tissue disorders) | 12 | 4 | 5 | 24 | 21 | 9
Back pain (Musculoskeletal and connective tissue disorders) | 8 | 6 | 12 | 19 | 24 | 28
Headache (Nervous system disorders) | 15 | 8 | 13 | 25 | 14 | 22
Pollakiuria (Renal and urinary disorders) | 6 | 6 | 12 | 10 | 11 | 15
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 8 | 18 | 13
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 16 | 11 | 13
Oedema peripheral (General disorders) | 0 | 0 | 0 | 17 | 6 | 2
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 8 | 15 | 11
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 13 | 9 | 6
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 0 | 0 | 1 | 13 | 11
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 19 | 6 | 6
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 13 | 4 | 6
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 11 | 16 | 11
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 13 | 9 | 6
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 6 | 5 | 12
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 22 | 17 | 18
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 15 | 11 | 7
Hypertension (Vascular disorders) | 0 | 0 | 0 | 12 | 5 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested in writing, such publication will be withheld for up to an additional 60 days.